CLINICAL TRIAL: NCT03599401
Title: Comparison of Effectiveness of Low Dose Aspirin Vs Omega 3 Fatty Acids as Adjuvants to Non-surgical Periodontal Therapy in Type II Diabetic Patients With Chronic Periodontitis
Brief Title: Effect of Aspirin Vs Omega 3 Fatty Acid After Scaling and Root Planing in Type II Diabetic Patients With Chronic Periodontitis
Acronym: EAOFASRPDMCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, Rampally Prathyusha, Student, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PERIO; D159206042 (Other: Dr. N T R UNIVERSITY OF HEALTH SCIENCES)
Record Dates: First submitted 2018-07-10; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Periodontitis; Type2 Diabetes
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: A total of 42 subjects participated in the study. All the subjects underwent scaling and root planning and were divided into 3 groups Group 1 - low dose aspirin ( 75 mg) once daily Group 2 - omega 3 fatty acids (500 mg) twice daily Group 3 - placebo once daily
Who Masked: Participant, Outcomes Assessor
Masking Description: Sealed Envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aspirin Group (Group I) (Active Comparator): 14 Patients in Group I underwent scaling and root planing using ultrasonic scalers after which 75 mgms of Aspirin was administered orally, once daily for 3 months
  Interventions: Other: Scaling and root planing
- Omega 3 Fatty acid Group (Group II) (Active Comparator): 14 Patients in Group II were given 500 mgms of Omega 3 Fatty Acid orally, twice daily for 3 months after scaling and root planing using ultrasonic scalers.
  Interventions: Other: Scaling and root planing
- Placebo Group (Group III) (Placebo Comparator): 14 Patients in Group III was given Placebo, which was administered orally, twice daily for 3 months after scaling and root planing using ultrasonic scalers.
  Interventions: Other: Scaling and root planing

INTERVENTIONS:
Other: Scaling and root planing — Scaling and root planing was done by using ultrasonic scalers with high speed suction apparatus to prevent aerosol contamination.
  .
  Other Names: Nonsurgical periodontal therapy

SUMMARY:
The main aim and objective of this study is to compare the effectiveness of low dose aspirin vs omega 3 fatty acids as adjuvants to non-surgical periodontal therapy and also to evaluate the levels of pentraxin 3 and glycosylated haemoglobin in diabetic patients with chronic periodontitis

DETAILED DESCRIPTION:
There is an established bi-directional relationship between diabetes mellitus and periodontitis. Periodontitis causes systemic inflammation by the entry of oral pathogens and their virulence factors that adversely affect diabetic control in terms of elevated HbA1c levels.

Host modulatory therapy (HMT) is a strategy prescribed as an adjunct to conventional periodontal treatment by downregulating inflammation and promoting protective or regenerative responses. Different drugs have been evaluated as HMT including NSAIDS, Doxycycline, Bisphosphonates.

Aspirin has the unique position as HMT drug. It inhibits prostanoid production and induces 15- epi- lipoxins which are bioactive than native lipoxins.

Omega 3 fatty acids including Docosahexaenoic acid and Eicosapentaenoic acid due to their anti-inflammatory, antithrombotic, hypolipidemia and vasodilator effect, reduce the inflammatory mediators to levels of healthy tissues.

Pentraxins(PTX3) are classic acute phase proteins. They are a superfamily of evolutionarily conserved proteins considered to be the markers of acute phase inflammation. PTX3 is also known as TNF stimulated gene. It is produced abundantly in periodontal tissue by neutrophils, fibroblasts, monocytes and epithelial cells. The plasma levels of PTX3 is raised in inflammatory conditions. Hence it is taken as a biomarker.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type II Diabetes
* Patients with Chronic periodontitis.
* Clinical attachment loss ≥ 4 mm
* Probing depths ≥ 5mm.
* 14 teeth should be present
* Diabetic patients having HbA1C levels ≥ 6%

Exclusion Criteria:

* Pregnant and lactating women
* Smokers
* Patients with any auto immune or systemic disorder other than type II Diabetes
* Use of Medicines or antibiotic 3 months before
* History of periodontal treatment within 12 months
* Suspected intolerance to Aspirin

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
Change in Plasma Pentraxin 3 levels | Base line and 3 months after scaling and root planning
  Blood samples were collected by venepuncture of anti-cubital vein. 1ml of blood was collected. 1ml blood was subjected to centrifugation at 3000rpm for 10 min. The supernatant straw colored fluid (plasma) was separated into storage vial for plasma pentraxin 3
Change in Glycosylated Hemoglobin levels | Base line and 3 months after scaling and root planning
  Blood samples were collected by venepuncture of anti-cubital vein. 1ml of blood was collected and was used for glycosylated hemoglobin (HbA1c) estimation

SECONDARY OUTCOMES:
Change in Gingival Index | Base line and 3 months after scaling and root planning
  The severity of gingivitis was scored on all surfaces of selected teeth with Williams periodontal probe.Index teeth- 16, 12, 24, 36, 32, 44 .
  CALCULATION:
  Score around each tooth was totaled and divided by 4- score of tooth Index score- total of all scores per tooth/no. of teeth examined Inference 0.1-1.0- mild gingivitis 1.1-2.0- moderate gingivitis 2.1- 3.0- severe gingivitis
Change in Pocket Probing Depth | Base line and 3 months after scaling and root planning
  The distance from the gingival margin to the base of the pocket was measured in millimeters using Williams periodontal probe
Change in Clinical attachment level | Base line and 3 months after scaling and root planning
  The distance from the cemento-enamel junction to the alveolar crest was measured in millimeters using Williams periodontal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Prathyusha Rampally, MDS, Principal Investigator — Panineeya Mahavidhyalaya Institute of Dental Sciences
Locations (1):
- Panineeya Mahavidhyalaya Institute of Dental Sciences, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elwakeel NM, Hazaa HH. Effect of omega 3 fatty acids plus low-dose aspirin on both clinical and biochemical profiles of patients with chronic periodontitis and type 2 diabetes: a randomized double blind placebo-controlled study. J Periodontal Res. 2015 Dec;50(6):721-9. doi: 10.1111/jre.12257. Epub 2015 Jan 21. PMID 25604769
- [Background] Pradeep AR, Kathariya R, Raghavendra NM, Sharma A. Levels of pentraxin-3 in gingival crevicular fluid and plasma in periodontal health and disease. J Periodontol. 2011 May;82(5):734-41. doi: 10.1902/jop.2010.100526. Epub 2010 Nov 16. PMID 21080790